CLINICAL TRIAL: NCT03662191
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, THREE-PERIOD, THREE-SEQUENCE, SINGLE-DOSE, CROSSOVER STUDY IN FASTED HEALTHY SUBJECTS, TO ASSESS THE SAFETY, PHARMACOKINETICS AND ORAL BIOAVAILABILITY OF TAFAMIDIS FREE ACID WET-MILLED SUSPENSION DOSES, RELATIVE TO 4 X 20 MG COMMERCIAL TAFAMIDIS MEGLUMINE CAPSULES
Brief Title: Phase I Safety, Pharmacokinetics and Bioavailability Study Comparing Rate and Extent of Absorption of Two Different Forms of Tafamidis (PF-6291826)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B3461059; 2017-004935-35 (EudraCT Number); BA STUDY (Other: Alias Study Number)
Record Dates: First submitted 2018-08-23; First posted 2018-09-07 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A (Experimental): 4 × 20 mg commercial tafamidis meglumine administered as soft gelatin capsules under fasted conditions
  Interventions: Drug: Tafamidis
- Treatment B (Experimental): 10 mgA tafamidis free acid administered as a wet-milled suspension under fasted conditions
  Interventions: Drug: Tafamidis
- Treatment C (Experimental): a dose of tafamidis free acid projected to be an equivalent of 4 × 20 mg commercial tafamidis meglumine administered as a wet-milled suspension under fasted conditions
  Interventions: Drug: Tafamidis
- Treatment D (Experimental): a dose of tafamidis free acid projected to be an equivalent of 5 × 20 mg commercial tafamidis meglumine administered as a wet-milled suspension under fasted conditions
  Interventions: Drug: Tafamidis

INTERVENTIONS:
Drug: Tafamidis — bioavailability study

SUMMARY:
2 different formulations and 4 different single doses of tafamidis will be compared. All subjects will receive both formulations and 3 different doses. Subjects will be fasted before taking the drug. After swallowing single dose of tafamidis, tafamidis blood concentrations will be measured periodically for 8 days. After another 16 days, all subjects will repeat the procedure twice, each time with the other formulation/dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females of non-child bearing potential.
* Body Mass Index (BMI) of 17.5 to 30.5 and total body weight more than 50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Blood pressure at screening visit of greater than 140 mm Hg (systolic) or 90 mg Hg (diastolic).
* Use of prescription or nonprescription drugs supplements within 7 days prior to the study.
* Fertile male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
1. Area under the plasma concentration-time profile from time 0 extrapolated to infinite time (AUCinf) | 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hrs
2. Maximum Observed Plasma Concentration (Cmax) | 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hrs

SECONDARY OUTCOMES:
1. Area under the plasma concentration-time profile from time 0 to 24 hours post-dose (AUC24) | 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hrs
2. Area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (AUClast) | 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hrs
3. Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3461059&StudyName=A+Phase+1%2C+Open-label%2C+Randomized%2C+Three-period%2C+Three-sequence%2C+Single-dose%2C+Crossover+Study+In+Fasted+Healthy+Subjects%2C+To+Assess+The+Safety%2C+Pharmacokinetics+And+Oral+Bioavailability+Of+Tafamidis+Free+Acid+Wet-milled+Suspension+Doses%2C+Relative+To+4+X+20+Mg+Commercial+Tafamidis+Meglumine+Capsules